CLINICAL TRIAL: NCT07139366
Title: Efficacy and Safety of Saccharomyces Boulardii Combined With Bismuth Quadruple Therapy for Helicobacter Pylori Rescue Treatment: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Saccharomyces Boulardii Combined With Bismuth Quadruple Therapy for Helicobacter Pylori Rescue Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yongquan Shi (Other)
Responsible Party: Sponsor-Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20252348-F-1
Record Dates: First submitted 2025-08-12; First posted 2025-08-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Gastritis; Dyspepsia; Helicobacter Pylori Infection; Gastric Cancer; Peptic Ulcer
MeSH Terms: conditions — Gastritis; Dyspepsia; Stomach Neoplasms; Peptic Ulcer | interventions — Bismuth; Esomeprazole; Tetracycline; Furazolidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saccharomyces boulardii combined with Bismuth-containing quadruple therapy (Experimental): Saccharomyces boulardii powder 500 mg twice daily for 14 days#Tetracycline 500mg three time daily for 14 days#furazolidone 100 mg, esomeprazole 20 mg, and Bismuth 220mg by mouth, twice daily for 14 days.
  Interventions: Drug: Bismuth; Drug: Esomeprazole; Drug: Tetracycline; Drug: Furazolidone; Drug: Saccharomyces Boulardii Oral Powder
- Bismuth-containing quadruple therapy (Active Comparator): Tetracycline 500mg three time daily for 14 days#furazolidone 100 mg, esomeprazole 20 mg, and Bismuth 220mg by mouth, twice daily for 14 days.
  Interventions: Drug: Bismuth; Drug: Esomeprazole; Drug: Tetracycline; Drug: Furazolidone

INTERVENTIONS:
Drug: Bismuth — Bismuth-containing quadruple therapy: given for 14 days at a dose of bismuth 110 mg 2 capsules BID plus esomeprazole 20 mg 1 tablets BID#tetracycline 250mg 2 capsules TID and furazolidone 100mg 1 tablets BID
Drug: Esomeprazole — Bismuth-containing quadruple therapy: given for 14 days at a dose of esomeprazole 20mg 1 tablets BID plus bismuth 110 mg 2 capsules BID#tetracycline 250mg 2 capsules TID and furazolidone 100mg 1 tablets BID
Drug: Tetracycline — Bismuth-containing quadruple therapy:given for 14 days at a dose of tetracycline 250mg 2 capsules TID plus furazolidone 100mg 1 tablets BID#esomeprazole 20 mg 1 tablets BID and bismuth 110 mg 2 capsules BID
Drug: Furazolidone — Bismuth-containing quadruple therapy:given for 14 days at a dose of furazolidone 100mg 1 tablets BID plus tetracycline 250mg 2 capsules TID#esomeprazole 20 mg 1 tablets BID and bismuth 110 mg 2 capsules BID
Drug: Saccharomyces Boulardii Oral Powder — Saccharomyces boulardii combined with Bismuth-containing quadruple therapy:given for 14 days at a dose of Saccharomyces boulardii powder 250 mg 2 packets BID#bismuth 110 mg 2 capsules BID plus esomeprazole 20 mg 1 tablets BID#tetracycline 250mg 2 capsules TID and furazolidone 100mg 1 tablets BID
  Arms: Saccharomyces boulardii combined with Bismuth-containing quadruple therapy

SUMMARY:
This study aims at evaluating efficacy and safety of Saccharomyces boulardii combined with bismuth-containing quadruple Therapy versus bismuth-containing quadruple Therapy(bismuth#esomeprazole#tetracycline and furazolidone) in H. pylori rescue therapy. It is hypothesized that Saccharomyces boulardii combined with bismuth-containing quadruple Therapy is superior to bismuth-containing quadruple Therapy. Patients with confirmed failure of H. pylori eradication will be randomized to one of the treatments described above. At week 6 follow-up visits, a urea breath test#rapid urease test or helicobacter pylori stool antigen test will be performed to confirm eradication.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up. Screening: this phase will last a maximum of 14 days and subjects eligibility will be evaluated after signing informed consent. One of urea breath test#rapid urease test or helicobacter pylori stool antigen test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects are randomly assigned to treatment and will be treated for 14 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 14 and 16.

Follow-up: includes one visits. Approximately 28 days after the end of treatment. Eradication of H. Pylori will be confirmed by one of urea breath test#rapid urease test or helicobacter pylori stool antigen test.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18~75, both gender.
* Patients who had failed H.pylori eradication therapies .
* Women are eligible if they are not pregnant or nursing, and if they are of childbearing potential they are required to use medically acceptable contraception for the duration of the study and 30 days thereafter.

Exclusion Criteria:

* Patients who have previously used tetracycline and furazolidone antibiotics to eradicate infection with H. pylori.
* Contraindications to study drugs.
* Substantial organ impairment, severe or unstable cardiopulmonary or endocrine disease.
* Constant use of anti-ulcer drugs ( including taking proton-pump.inhibitors(PPI) within 2 weeks before the [13C] urea breath test), antibiotics or bismuth complexes (more than 3 times /1 month before screening).
* Pregnant or lactating women.
* Underwent upper gastrointestinal Surgery.
* Dysphagia.
* Evidence of bleeding or iron efficiency anemia.
* A history of malignancy.
* Drug or alcohol abuse history in the past 1 year.
* Systemic use of corticosteroids, non steroidal anti-inflammatory drugs, anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
* Mental disorder.
* Enrolled in other clinical trials in the past 3 months.
* Refuse to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1248 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | 28 days after treatment
  The primary end point of this study is H.pylori eradication#established by negative [13C] urea breath test #DOB value below 3.9#28 days after the end of eradication

SECONDARY OUTCOMES:
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache,dizziness,skin rash,other gastrointestinal disorders,pyrexia,cough and back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No